CLINICAL TRIAL: NCT07194525
Title: Feasibility and Safety of an Ileus Management Protocol for Postoperative Ileus
Brief Title: Feasibility and Safety of an Ileus Management Protocol for Postoperative Ileus After Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, David Fuks, Professor, Head of the Department of Visceral surgery, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-00759
Record Dates: First submitted 2025-09-11; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Ileus Postoperative; Nasogastric Tube
Keywords: ileus postoperative; treatment algorithm; hospital stay
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ileus Management Protocol (I-MAP) (Other): All enrolled patients who develop postoperative ileus after abdominal surgery are managed according to the standardized Ileus Management Protocol (I-MAP). The algorithm is based on nasogastric tube (NGT) output and includes stepwise interventions:
  Administration of water-soluble contrast (Telebrix® gastro, ioxitalamic acid 300 mg/mL) via NGT, followed by a clamp test at 4 hours.
  Diagnostic imaging (CT-scan or X-ray) if ileus persists or small bowel obstruction is suspected.
  Intravenous Neostigmine® (2.5 mg in 500 mL NaCl 0.9% over 5 hours) as a prokinetic, only after small bowel obstruction is excluded.
  The protocol is applied until resolution of postoperative ileus or requirement for further intervention.
  Interventions: Other: A standardized treatment algorithm for postoperative ileus after abdominal surgery, based on nasogastric tube output and including stepwise use of water-soluble contrast, imaging, and prokinetic medic

INTERVENTIONS:
Other: A standardized treatment algorithm for postoperative ileus after abdominal surgery, based on nasogastric tube output and including stepwise use of water-soluble contrast, imaging, and prokinetic medic — The Ileus Management Protocol (I-MAP) is a standardized algorithm for the treatment of postoperative ileus (POI) after abdominal surgery. Management decisions are based on nasogastric tube (NGT) output measured every 12 hours. Depending on output and tolerance, patients may receive:
  Water-soluble contrast (Telebrix® gastro, ioxitalamic acid 300 mg/mL) administered via NGT, followed by a clamp test at 4 hours.
  Diagnostic imaging (CT-scan or X-ray) if ileus persists or small bowel obstruction is suspected.
  Intravenous Neostigmine® (2.5 mg diluted in 500 mL NaCl 0.9%, infused over 5 hours) as a prokinetic, only after small bowel obstruction is excluded.
  The protocol is applied until resolution of POI or requirement of further intervention.

SUMMARY:
The goal of this clinical trial is to evaluate whether a standardized treatment algorithm, the Ileus Management Protocol (I-MAP), is feasible and safe for the management of patients who develop postoperative ileus (POI) within 30 days after abdominal surgery.

The main questions it aims to answer are:

Can I-MAP be applied consistently, with ≥85% adherence, in eligible patients with POI?

Is the use of I-MAP associated with acceptable safety outcomes, including low rates of complications such as pneumonia, aspiration, and adverse events?

This study does not include a comparison group. All participants are assigned to the I-MAP protocol, and outcomes are evaluated prospectively.

Participants will:

Be monitored for POI symptoms (nausea, vomiting, bloating, absence of gas/stool).

Receive standardized management according to I-MAP, which includes:

Daily assessment of nasogastric tube (NGT) output.

Water-soluble contrast administration via NGT when indicated.

Imaging (CT scan or X-ray) if obstruction is suspected.

Neostigmine administration if small bowel obstruction is excluded.

The primary endpoint is the feasibility of I-MAP, defined as the proportion of POI patients treated according to the algorithm. Secondary outcomes include NGT reinsertion, duration of NGT placement, hospital length of stay, conservative treatment failure, and complications related to POI.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age.
* Patients who undergo abdominal surgery and develop postoperative ileus (POI) within 30 days.
* Provided general consent for participation.

Exclusion Criteria:

* Preoperative bowel obstruction.
* Anastomotic leak.
* Prophylactic nasogastric tube (NGT) placement.
* Pregnancy.
* Lack of general consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of the I-MAP Algorithm | From surgery until resolution of postoperative ileus (up to 30 days).
  Proportion of eligible patients with postoperative ileus who are managed according to the standardized Ileus Management Protocol (I-MAP). A protocol adherence rate of ≥85% is considered indicative of feasibility.

SECONDARY OUTCOMES:
Nasogastric Tube (NGT) Reinsertion | From surgery until resolution of postoperative ileus (up to 30 days).
  Number and proportion of patients requiring reinsertion of the nasogastric tube after initial removal.
Duration of Nasogastric Tube Placement | From initial placement until final removal, during index hospital stay, up to 30 days.
  Total number of days the nasogastric tube remained in place for each patient.
Hospital Length of Stay (LOS) | From day of surgery until discharge, up to 30 days.
  Total number of days spent in hospital after surgery, including any delays related to postoperative ileus management.
Conservative Treatment Failure | From initiation of conservative treatment until resolution of ileus or re-intervention, up to 30 days after surgery.
  Proportion of patients in whom conservative management per I-MAP failed, requiring additional interventions
Postoperative Ileus-Related Complications | From initiation of conservative treatment until resolution of ileus, up to 30 days after surgery.
  Incidence of complications potentially related to postoperative ileus, including pneumonia, bronchoaspiration, and other adverse events associated with POI management.

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Grass, MD, Study Director — University of Lausanne Hospitals; David Fuks, MD, Study Chair — University of Lausanne Hospitals; Teresa Torres, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Centre hospitalier universitaire vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-07-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT07194525/Prot_000.pdf